CLINICAL TRIAL: NCT02220062
Title: Randomized, Controlled Trial of Endoscopic Ultrasound-Guided Bilateral Celiac Plexus Neurolysis vs Celiac Ganglia Neurolysis to Control Pain in Inoperable Pancreatic Cancer Patients With Inadequate Pain Control by Pain Killer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Kyun Lee, Professor, Department of Gastroenterology, Sungkyunkwan University School of Medicine, Samsung Medical center, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-02-088-005
Record Dates: First submitted 2014-07-21; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- EUS-CPN group (Active Comparator): Group that be performed by Endoscopic ultrasound guided bilateral celiac plexus neurolysis
  Interventions: Procedure: EUS-CPN
- EUS-CGN group (Experimental): Group that be performed by Endoscopic ultrasound guided celiac ganglia neurolysis
  Interventions: Procedure: EUS-CGN

INTERVENTIONS:
Procedure: EUS-CPN — After initially identifying the celiac trunk on endoscopic ultrasound, each injection of 5~10cc ethanol would be performed as bilateral injections at the celiac trunk.
  Arms: EUS-CPN group
Procedure: EUS-CGN — First, identify celiac ganglia. If the celiac ganglia are visualized under linear EUS, the injection of 2~3cc ethanol are applied directly into the each ganglia. If the ganglia are not identified by EUS, bilateral EUS-CPN would be performed
  Arms: EUS-CGN group

SUMMARY:
Pancreatic cancer related pain can be difficult to control, even with high doses of narcotics, whose adverse effects may further impair quality of life. So EUS-CPN(endoscopic ultrasound guided celiac plexus neurolysis) is well established as an effective technique for controlling pain and reducing narcotic requirements in patients with pancreatic cancer. Recently, celiac ganglia can be visualized and accessed by endoscopic ultrasound. So it allows for direct injection into individual celiac ganglia to perform celiac ganglia neurolysis. This more precise delivery of therapeutic drug will offers the potential for enhanced efficacy and safety. To evaluate this hypothesis, this randomized controlled trial aimed to compare the efficacy and safety of EUS-CGN(Endoscopic ultrasound guided celiac ganglia neurolysis) vs. Bilateral EUS-CPN(Endoscopic ultrasound guided celiac plexus neurolysis) in providing relief from pancreas cancer-related pain.

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years old age (above 70 years old age, need the consent of the legal representative)
2. Inoperable pancreatic cancer patients
3. Pancreatic cancer patients with inadequate pain control by pain killer (VAS score 4 points or more)
4. Patient who agree to participate in this study

Exclusion Criteria:

1. Abnormal clotting (international normalized ratio ≥1.5)
2. Reduced platelet count (≤50000/μL)
3. Use of anticoagulation agents
4. Presence of gastric and/or esophageal varices
5. Anatomical deformity due to past surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
percentage of participants with 50% decrease or less than 3 points in Pain Visual Analogue Scale (VAS) | 1 week after procedure